CLINICAL TRIAL: NCT01552447
Title: A Multi-center Randomized Controlled Clinical Trial Evaluating Two Application Regimens of Human Amniotic Membrane Grafting and Standard of Care Versus Standard of Care Alone in the Treatment of Venous Leg Ulcers.
Brief Title: Human Amniotic Membrane Grafting and Standard of Care Versus Standard of Care Alone in the Treatment of Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFVLU001
Record Dates: First submitted 2012-03-06; First posted 2012-03-13 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 application of EpiFix (Other): 1 x dehydrated human amnion/chorion membrane
  Interventions: Other: EpiFix; Other: Compression Therapy
- 2 applications of EpiFix (Other): 2 x dehydrated human amnion/chorion membrane
  Interventions: Other: EpiFix; Other: Compression Therapy
- Standard of care (Other): Compression bandaging
  Interventions: Other: Compression Therapy

INTERVENTIONS:
Other: EpiFix — Dehydrated placental tissue
  Arms: 1 application of EpiFix; 2 applications of EpiFix
Other: Compression Therapy — Compression bandaging

SUMMARY:
The purpose of this study is to determine whether the EpiFix human amniotic membrane is effective in the treatment of venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Ankle Brachial Pressure Index (ABI) > 0.75
* Presence of a venous leg ulcer extending through the full thickness of the skin but not down to muscle, tendon or bone
* Study ulcer has been present for at least one month prior to the initial screening visit, and is excluded if it has undergone 12 months of continuous high strength compression therapy over its duration
* Study ulcer is a minimum of 2 cm2 and a maximum of 20 cm2 at the Randomization visit
* The target ulcer has been treated with compression therapy for at least 14 days prior to randomization
* Ulcer has a clean, granulating base with minimal adherent slough at the Randomization visit
* Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
* Patient understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen
* Patient has read and signed the IRB/IEC approved Informed Consent Form before screening procedures are undertaken

Exclusion Criteria:

* Study ulcer(s) deemed by the investigator to be caused by a medical condition other than venous insufficiency
* Study ulcer exhibits clinical signs and symptoms of infection.
* Non-mobile i.e. not ambulatory, or bed ridden
* Study ulcer, in the opinion of the investigator, is suspicious for cancer should undergo an ulcer biopsy to rule out a carcinoma of the ulcer
* Patients with a history of more than two weeks treatment with immuno-suppressants (including systemic corticosteroids), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to initial screening, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study
* Patients on any investigational drug(s) or therapeutic device(s) within 30 days preceding Screening
* History of radiation at the ulcer site
* Known history of having Acquired Immunodeficiency Syndrome (AIDS) or HIV.
* Study ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days
* Study ulcer requiring negative pressure wound therapy or hyperbaric oxygen during the course of the trial.
* Patients who are unable to understand the aims and objectives of the trial
* Presence of any condition(s) which seriously compromises the subject's ability to complete this study, or has a known history of poor adherence with medical treatment
* NYHA Class III and IV congestive heart failure (CHF), as defined by the following criteria: Class III: Symptoms with moderate exertion; Class IV: Symptoms at rest
* Ulcers on the dorsum of the foot or with more than 50% of the ulcer below the malleolus are excluded.
* Pregnant or breast feeding
* Currently taking medications which could affect graft incorporation.(supervising physicians discretion)
* Allergic to gentamicin and streptomycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The proportion of wounds achieving 40% closure in patients treated with amniotic membrane vs. standard of care | 4 week

SECONDARY OUTCOMES:
The proportion of wounds achieving 40% closure in patients treated with one application of amniotic membrane vs. standard of care | 4 week
The proportion of wounds achieving 40% closure in patients treated with one application of amniotic membrane vs. 2 applications of amniotic membrane | 4 week
The proportion of wounds achieving 40% closure in patients treated with two applications of amniotic membrane vs. standard of care | 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD, Principal Investigator — Penn North Centers for Advanced Wound Care
Locations (5):
- United States (5):
  - Eric J. Lullove DPM, Boca Raton, Florida
  - MetroWest Medical Center, Framingham, Massachusetts
  - St. Johns Wound Center, Tulsa, Oklahoma
  - St. Vincent's Health Center, Erie, Pennsylvania
  - Armstrong County Memorial Hospital, Kittanning, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided